CLINICAL TRIAL: NCT02142608
Title: A Pilot Clinical Trial Using BR55 Ultrasound Contrast Agent in the Assessment of Prostate Cancer by Molecular Imaging of VEGFR2
Brief Title: A Pilot Trial Using BR55 Ultrasound Contrast Agent in the Assessment of Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BR55-105
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Ultrasound Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BR55 (Experimental): All patients received BR55 as a single intravenous injection at the dose of 0.03 mL/kg...
  Interventions: Drug: BR55

INTERVENTIONS:
Drug: BR55 — Ultrasound contrast agent

SUMMARY:
Pilot study to evaluate the ability of BR55 to identify prostate cancer lesions with Gleason Score ≥7 by ultrasound molecular imaging on the basis of a visual score in comparison with histopathology results

DETAILED DESCRIPTION:
This multi-centre, open label, prospective, pilot study was designed to assess the ability of BR55 to detect VEGFR2 in human prostate cancer by Ultrasound Molecular Imaging (USMI). The binding of BR55 to VEGFR2 (focal enhancement still visible after significant decrease in signal from circulating microbubbles seen) was assessed at USMI and VEGFR2 expression was to be confirmed by immunohistochemistry (IHC) analysis including VEGFR2 and CD31 staining.

ELIGIBILITY:
Inclusion Criteria:

* Male, age between 50-70 years old
* Increased Prostate-Specific Antigen (PSA) level >4 ng/mL
* Known prostate cancer
* Scheduled for prostatectomy not earlier than 3 days and not later than 30 days following BR55 administration (with the exception of training cases where this requirement is not applicable)
* Provided written informed consent and willing to comply with protocol requirements

Exclusion Criteria:

* Documented acute prostatitis or urinary tract infections
* Known to suffer from stable angina pectoris and/or proven coronary disease, or have symptoms suspicious of coronary disease
* History of any clinically unstable cardiac condition including class III/IV cardiac failure or right-to left shunts
* Severe cardiac rhythm disorders within the last 7 days
* Severe pulmonary hypertension or uncontrolled systemic hypertension or respiratory distress syndrome
* Received a prostate biopsy procedure within 30 days before admission into the study
* Determined by investigator to be clinically unsuitable for the study
* Participated in a concurrent clinical trial or has participated in another clinical trial with an investigational compound within the past 30 days

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luigia Storto, M.D., Study Director — Bracco Diagnostics, Inc
Locations (2):
- Translational Molecular Imaging Lab, Stanford, California, United States
- Service d'Imagerie Diagnostique et Interventionnelle de l'Adulte, Bordeaux, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 patients were recruited, but only 18 were dosed. Of the 18 dosed, 4 were training cases evaluated for safety only. Of the remaining 14 patients, 1 had no evaluable images; therefore, only 13 patients were included in the Efficacy Population.
Pre-assignment Details: One participant was not dosed with BR55.
  Patient signed informed consent but did not receive investigational product. During pre-dose safety evaluations, it was discovered that patient may have potentially clinical significant abnormal ECGs (atrial fibrillation).
Period: Overall Study
Arm/Group | BR55
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BR55
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (4.68)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 12
  >= 65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Black | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 16
  Other | 0
Weight [Mean (Standard Deviation); unit: kg] | 83.62 (15.573)
Height [Mean (Standard Deviation); unit: cm] | 172.6 (8.71)

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions With Gleason Score ≥ 7 Identified by Ultrasound Molecular Imaging
Description: To assess the ability of BR55 to identify prostate cancer lesions with a Gleason score ≥ 7 using histopathology as truth standard
Time Frame: Within 30 minutes after administration of BR55
Population: BR55 binding level versus Gleason score in malignant lesions from off-site histopathology
Measure: Number; unit: number of lesions
Groups:
- BR55: Ultrasound Image Assessment
Arm/Group | BR55
Number analyzed (Participants) | 13
number of lesions
  Gleason score ≥7 | 17
  With binding | 8

2. Secondary Outcome: Number of Participants With Adverse Events
Description: To obtain safety data in subjects administered BR55
Time Frame: 24 hours post-dose
Measure: Number; unit: participants
Arm/Group | BR55
Number analyzed (Participants) | 18
participants
  Number of subjects with AEs | 1
  Number of subjects with AEs by intensity - Mild | 1
  Number of subjects with AEs by intensity -Moderate | 0
  Number of subjects with AEs by intensity - Severe | 0
  Number of subjects with serious AEs | 0
  Number of subjects who discontinued due to AEs | 0
  Number of deaths | 0

ADVERSE EVENTS:
Time Frame: All adverse events that occurred from the time the patient signed the Informed Consent Form until 24 hours after the last administration of BR55 were recorded.
Arm/Group | BR55
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BR55 (N=18)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No